CLINICAL TRIAL: NCT06223087
Title: Effects of Winter Swimming on Blood Morphological, Rheological, and Biochemical Indicators and Oxidative Stress in Males
Brief Title: Effects of Winter Swimming on Blood Indicators and Oxidative Stress in Males
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Principal Investigator, Aneta Teleglow, Head of Blood Physiology Laboratory, University School of Physical Education, Krakow, Poland
Other Study IDs: 296/BS/INP/2021
Record Dates: First submitted 2023-12-30; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Cold Exposure
Keywords: blood; rheology; cold; blood morphology; biochemistry; exercise
MeSH Terms: conditions — Common Cold; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: group not practicing winter swimming
- winter swimmers: group practicing winter swimming
  Interventions: Other: winter swimming

INTERVENTIONS:
Other: winter swimming — Intervention involves bathing/swimming in cold water during the winter months in open waters
  Groups: winter swimmers

SUMMARY:
Exposure of the human body to cold water triggers numerous beneficial physiological changes. The study aimed to assess the impact of regular winter swimming on blood morphological, rheological, and biochemical indicators and activity of antioxidant enzymes in males. The study includes winter swimmers and a control group. Blood samples were taken twice - before the start (November) of the winter swimming season and after its end (March). The average duration of ice water baths was 3-5 minutes, with a minimum frequency of once a week. The water temperature during the swimming did not exceed 10°C, approaching 0°C during the winter period.

ELIGIBILITY:
Inclusion Criteria:

* Good health, practitioners of winter swimming
* control group: never did winter swimming and had a sedentary lifestyle.

Exclusion Criteria:

* medical contraindications to winter bathing

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Experienced in winter swimming, regularly swimming in cold water (open water) at least once a week in the period November - March
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
blood sampling: platelets and leukocytes | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Measurements of:
  Platelets [thousands/μl], Leukocytes [thousands/μl], Neutrophils [thousands/μl], Eosinophils [thousands/μl], Basophils [thousands/μl], Lymphocytes [thousands/μl], Monocytes [thousands/μl].
blood sampling: erythrocytes | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Measurement of:
  Erythrocytes [mln/μl],
blood sampling: haemoglobin | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of:
  Haemoglobin [g/dl], mean corpuscular haemoglobin concentration (MCHC) [g/dl],
blood sampling: haematocrit | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of:
  haematocrit [%], red blood cell distribution width coefficient of variation (RDW-CV) [%],
blood sampling: haemoglobin mass | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of:
  mean corpuscular haemoglobin (MCH) [pg],
blood sampling: Erythrocytes | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of mean corpuscular volume (MCV) [fl], red blood cell distribution width standard deviation (RDW-SD) [fl],
blood sampling: rheology part 1 | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of red cell elongation index (EI) [arbitrary unit: AU], erythrocyte aggregation amplitude (AMP) [AU],
blood sampling: rheology part 2 | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of:
  aggregation index (AI) [%],
blood sampling:rheology part 3 | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of:
  half-time of total aggregation (t1/2) [s].
blood sampling: oxidative stress | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Measurement of catalase (CAT) [nmol/min/ml], and glutathione peroxidase (GPx) [nmol/min/ml].
blood sampling: oxidative stress - superoxide dismutase | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Measurement of superoxide dismutase (SOD) [U/ml],
blood biochemistry: Urea | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Measurement of:
  Urea [mmol/l].
blood sampling: Testosterone | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of Testosterone concentration [ng/dl],
blood sampling: Cortisol | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of Cortisol concentration [µg/dl],
blood biochemistry: Creatine | twice: before the start of cold swimming in November and 5 months later (March), after the end of winter swimming
  Determination of Creatinine concentration [µmol/l],

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Teleglow, Principal Investigator — University of Physical Education, Kraków, Poland
Locations (1):
- University of Physical Education, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teleglow A, Konieczny K, Dobija I, Kusmierczyk J, Tota L, Rembiasz K, Maciejczyk M. Effect of regular winter swimming on blood morphological, rheological, and biochemical indicators and activity of antioxidant enzymes in males. BMC Sports Sci Med Rehabil. 2024 Jun 21;16(1):138. doi: 10.1186/s13102-024-00932-3. PMID 38907310